CLINICAL TRIAL: NCT07038174
Title: A Study for Development and Testing of Fertility Preservation Decision Aid for Young Cancer Patients
Brief Title: A Study to Evaluate the Effectiveness of a Web-based Tool for Fertility Preservation in Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCC2024-0050
Record Dates: First submitted 2025-06-11; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Female; Neoplasms
MeSH Terms: conditions — Infertility, Female; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Received only the planned cancer treatment without any additional intervention
- Fertility preservation decision aid intervention group (Experimental): Visited the website containing the web-based decision aid regarding fertility preservation at least once before cancer treatment initiation to independently use the tool in a private setting
  Interventions: Other: Fertility preservation decision aid intervention group

INTERVENTIONS:
Other: Fertility preservation decision aid intervention group — Visited the website containing the web-based decision aid regarding fertility preservation at least once before cancer treatment initiation to independently use the tool in a private setting
  Arms: Fertility preservation decision aid intervention group

SUMMARY:
[Background] The number of young cancer patients is increasing, and they may experience impairment or loss of reproductive function due to cancer treatments such as surgery, radiation therapy, and chemotherapy.

Although various medical methods to preserve fertility have been developed, due to the complexity and medical specialization of these methods, there is an urgent need to support understanding and decision-making regarding these options in clinical practice.

While referrals to fertility specialists for counseling are possible, most young cancer patients do not receive such consultations before treatment. Even those who do often report decisional conflict due to confusion about the information and difficulty in reflecting personal values in the decision-making process.

Although decision aids have been developed in other countries, cultural, linguistic, and healthcare system differences make it difficult to apply these tools in Korea.

Therefore, there is a need to develop a decision aid tailored to female cancer patients in Korea for use in local clinical settings to support fertility preservation decisions.

[Study Objective] To develop a web-based decision aid and evaluate its impact on decisional conflict, fertility preservation-related knowledge, decision self-efficacy, depression, and quality of life, in order to assess the effectiveness of the decision aid.

[Study Hypothesis]

The use of a web-based decision aid for fertility preservation will:

Reduce decisional conflict experienced by cancer patients during the decision-making process; Improve fertility preservation-related knowledge and decision self-efficacy; Reduce levels of depression and improve quality of life.

[Study Plan]

1. Study Design

   * Randomized clinical study
   * Prospective study
   * Two-arm randomized controlled trial (RCT)

     2. Study Method Female cancer patients visiting the outpatient clinic of the National Cancer Center will be screened to determine eligibility based on inclusion and exclusion criteria.

Patients who meet the criteria and voluntarily agree to participate will be enrolled in the study.

Participants will be randomly assigned to either the intervention group (who will use the decision aid) or the control group (who will receive standard cancer treatment as planned at the Cancer Center without any special tools).

The decision aid will be provided to the intervention group immediately after randomization. The control group will not receive any additional tools.

Outcomes will be measured at three time points for the intervention group: before the intervention (T0), one week after the intervention (T1), and one month after the intervention (T2).

For the control group, measurements will be taken at the same time points: immediately after randomization (T0), one week later (T1), and one month later (T2).

ELIGIBILITY:
Inclusion Criteria:

* Female cancer patients aged 18 to 40 who received treatment at the National Cancer Center between June 2025 and December 2025
* Voluntarily agreed to participate in the study
* Able to read, write, and communicate in Korean without difficulty

Exclusion Criteria:

* Patients who had already lost fertility prior to participating in the study
* Patients who had already undergone, or were scheduled to undergo, a specific fertility preservation procedure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict score | Before the intervention, one week after the intervention, and one month after the intervention.
  Name of the measurement: Decisional conflict score assessed by the Decisional Conflict Scale (DCS)
  Measurement tool: The Decisional Conflict Scale (DCS) - low literacy version Measure description: The level of decisional conflict experienced by participants regarding a health-related decision will be assessed using the Decisional Conflict Scale (DCS) - low literacy version, a validated 10-item questionnaire. Each item is rated on yes(0), unsure(2), no(4), and scores are converted to a 0-100 scale, with higher scores indicating greater decisional conflict. The unit of measure will be the mean total score on the DCS at the specified timepoint. Subscale scores (e.g., uncertainty, informed, values clarity, support, and effective decision) may also be calculated.
  Unit of measure: Mean scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict)

SECONDARY OUTCOMES:
Knowledge about fertility preservation | Before the intervention, one week after the intervention, and one month after the intervention.
  Name of the measurement: Knowledge about fertility preservation Measurement tool: Questionnaire developed by researchers Measure description: Knowledge about fertility preservation will be assessed using a questionnaire developed by researchers. To develop the questionnaire items, guidelines and prior studies on the development and evaluation of fertility preservation decision aids will be reviewed to extract essential and frequently asked information for cancer patients. A panel of experts will be consulted to evaluate the relevance of each item. After item selection, researchers will develop corresponding questions and response options, which will be reviewed and revised based on expert feedback.
  The measurement tool will be a customized questionnaire assessing FP knowledge, and the unit of measure will be the percentage of participants who answer each knowledge item correctly.
  Unit of measure: % of participants with correct answers (per item)
Depression severity | Before the intervention, one week after the intervention, and one month after the intervention.
  Name of the measurement: Depression severity assessed by the Patient Health Questionnaire-9 (PHQ-9) Measurement tool: Patient Health Questionnaire-9 (PHQ-9) Measure description: Depression severity will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a validated 9-item self-report questionnaire widely used to screen for and measure the severity of depressive symptoms. Each of the 9 items is scored on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater severity of depression. The unit of measure will be the mean total PHQ-9 score at each time point. Depression severity levels based on PHQ-9 score will be categorized as follows: 0-4: Minimal or no depression/5-9: Mild depression/10-14: Moderate depression/15-19: Moderately severe depression/20-27: Severe depression
  Unit of measure: Mean PHQ-9 total score (range: 0-27; higher scores = worse outcome)
Health-Related Quality of Life | Before the intervention, one week after the intervention, and one month after the intervention.
  Name of the measurement: Health-Related Quality of life assessed by the EuroQol 5-dimension 5-level (EQ-5D-5L) Measurement tool: EuroQol 5-dimension 5-level (EQ-5D-5L) Measure description: Health-related quality of life will be assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) instrument, a standardized and validated questionnaire developed by the EuroQol Group. The EQ-5D-5L evaluates five dimensions of health: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression Each dimension is rated on 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses generate a health profile that is converted into a utility index score based on a population-specific value set. The units of measure is EQ-5D-5L index score (range from <0 [worse than death] to 1 [full health])
  Unit of measure: Mean EQ-5D-5L index score (from 0 [worse than death] to 1 [full health])
Decision-Making Confidence | Before the intervention, one week after the intervention, and one month after the intervention.
  Name of the measurement: Decision-Making Confidence Assessed by the Decision Self-Efficacy Scale Measurement tool: Decision self-efficacy scale Measure description: Confidence in decision-making will be assessed using the Decision Self-Efficacy Scale, a validated 11-item questionnaire developed to measure individuals' self-confidence in engaging in health-related decision-making. Each item is rated on a 5-point Likert scale ranging from 0 (not at all confident) to 4 (very confident). The total raw score (0-44) is converted to a standardized score ranging from 0 to 100, where higher scores indicate greater decision-making self-efficacy. The scale assesses perceived ability to ask questions, express opinions, evaluate options, and participate in decisions about one's health care.
  Unit of measure: Mean score (0-100); higher = better decision-making self-efficacy
Counselling on fertility preservation | one month after the intervention
  Name of the measurement: Counseling on fertility preservation Measurement tool: Study-developed question (investigator-designed, not previously validated) Measure description:This outcome will assess whether participants received any counseling regarding fertility preservation after participation in the clinical trial. A validated measurement tool will not be used; instead, participants will be asked a direct yes/no question about whether they were counseled on fertility preservation options (e.g., egg or embryo freezing, ovarian tissue preservation) by a healthcare provider.
  Unit of measure: % of participants reporting receipt of counseling
Decision-making about fertility preservation | one month after the intervention
  Name of the measurement: Decision-making about fertility preservation Measurement tool: Study-developed question (investigator-designed, not previously validated) Measure description: This outcome assesses whether participants have made an actual decision regarding fertility preservation after participation in the clinical trial. A study-developed question will be used to ask participants directly whether they have decided to undergo fertility preservation procedures (such as egg freezing, embryo freezing, or ovarian tissue preservation) or have decided against it.
  The measurement tool is a study-specific, investigator-developed yes/no question, not based on a previously validated instrument.
  Unit of measure: % of participants reporting receipt of counseling
Readiness for decision-making | one week after the intervention
  Name of the measurement: Readiness for decision-making assessed by the Preparation for Decision-Making Scale Measurement tool: Preparation for Decision-Making Scale Measure description: Readiness for decision-making will be evaluated using the Preparation for Decision-Making Scale (PrepDM Scale), a validated questionnaire designed to assess how well individuals feel prepared to make health-related decisions after receiving information or decision support. The scale consists of 10 items, each rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (a great deal). The total score is calculated by summing item scores, then converted to a standardized score ranging from 0 to 100, where higher scores indicate greater perceived preparedness for decision-making. The unit of measure will be the mean PrepDM score (0-100).
  Unit of measure: Mean score (0-100); higher = better preparation for decision-making

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to concerns about participant privacy and the potential risk of re-identification, especially given the sensitive nature of the data. In addition, there are no current resources or infrastructure in place to support secure data sharing.

REFERENCES:
- [Derived] Jang J, Lee EM, Chung YK, Lee DO, Park HJ, Yim GW, Lee KS, Kim JH, Ko AR, Hong JH, Kang S. Development and pilot testing of a personalised decision aid for decision-making regarding fertility preservation in young female patients with cancer: a study protocol. BMJ Open. 2025 Aug 12;15(8):e090759. doi: 10.1136/bmjopen-2024-090759. PMID 40803737